CLINICAL TRIAL: NCT00704925
Title: Treatment of Lambert-Eaton Syndrome With 3, 4-Diaminopyridine
Brief Title: Treatment of Lambert-Eaton Syndrome With 3,4 DAP
Status: No longer available | Type: Expanded Access
Sponsor: David P. Richman, MD (Other)
Collaborators: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, David P. Richman, MD, Principal Investigator, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Other Study IDs: 200311036
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Lambert Eaton Myasthenic Syndrome
Keywords: Lambert Eaton Myasthenic Syndrome; 3,4 DAP; 3,4 Diaminopyridine
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

INTERVENTIONS:
Drug: 3, 4 DAP — Patients with clinically-confirmed LEMS will receive 3, 4 DAP by mouth in slowly increasing doses. Treatment will begin with 5 mg three times a day and will increase by 50% every two weeks to 10-15 mg three to six times a day, as clinically needed, and if tolerated.
  Other Names: 3,4 diaminopyridine

SUMMARY:
A new drug called 3,4-Diaminopyridine (3,4-DAP) is currently under investigation for treatment of the symptoms of Lambert-Eaton Myasthenic Syndrome (LEMS). This is an expanded access trial, which means that although data from this study will be collected and reported to the US Food and Drug Administration (FDA)and the drug manufacturer, this is not a formal study of drug in LEMS.

If you decide volunteer, you will be evaluated by a neurologist to determine your eligibility to receive 3, 4-DAP by a review of your medical history, medication regimen (the medications you are taking) and a neurological examination. If you are a female of child-bearing potential, a serum pregnancy test will be done to ensure that you are not pregnant. Once it is determined that this treatment is appropriate for your care, you will begin taking 3, 4 DAP by mouth in slowly increasing doses. Treatment will begin with 5mg three times a day, as clinically needed, and if tolerated. You will be monitored for strength and side effects by routine clinic visits at initial intervals of once a month, increasing to intervals of every 12 months as permitted. Blood will be drawn (approximately 1 tablespoon) at every clinic visit or as often as the investigator deems necessary to assess your liver/kidney function and blood counts. You will have an EKG (a test to see how your heart is functioning) at your first study visit, after 6 months of taking 3,4 DAP and again every 2 years. Treatment will be continued indefinitely if a good clinical response is achieved. This study is planned to last indefinitely.

The dosage of 3, 4DAP is individually adjusted. The usual range is 10-15 mg 3-4 times per day for the full effect and will increase by 50% every two weeks to 10-15 mg three to six times a day, as needed and if tolerated. Dosages above the full effect level will not provide an additional benefit and should not be used. 3, 4 DAP is a convulsant (causes seizures). A total of 100 mg/day is the maximum dosage allowed.

DETAILED DESCRIPTION:
Patients with clinically-confirmed LEMS will receive 3, 4-DAP by mouth in slowly increasing doses. Treatment will begin with 5 mg, three times a day and will increase by 50% every two weeks to 10-15 mg, three to six times a day, as clinically needed, and if tolerated. Patients will be monitored for strength and side effects via routine out-patient clinic visits at initial intervals of 1 month, increasing to intervals of 12 months as permitted. Results of treatment and adverse events will be reported to the FDA. Treatment will be continued indefinitely if a good clinical response is achieved and side effects are tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older, diagnosed with LEMS
* If female, have negative pregnancy test and if premenopausal, be willing to practice an effective form of birth control during the study.

Exclusion Criteria:

* Is known to have a sensitivity to 3, 4 DAP
* Has a history of past or current seizures
* Has a history of past or current severe asthma
* Is believed by the investigator to be unable to comply with the protocol
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: David Richman, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States